CLINICAL TRIAL: NCT05268458
Title: Myocarditis After SARS-CoV2-Vaccination: An International Patient Registry on Clinical Manifestations and Outcomes
Brief Title: Myocarditis After SARS-CoV2-Vaccination
Acronym: MYOVACC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Theresien Hospital Mannheim (Other)
Collaborators: University Hospital Heidelberg, GER (Unknown); GRN Hospital Weinheim, GER (Unknown); McGill University Health Care Montreal, CA (Unknown); Foothills Medical Centre Calgary, CA (Unknown); Sunnybrooks Research Institute Toronto, CA (Unknown); Unity Health St. Michael's Hospital Toronto, CA (Unknown)
Responsible Party: Principal Investigator, Marco Ochs, Attending, Cardiologist, Theresien Hospital Mannheim
Other Study IDs: TKH-032022-001
Record Dates: First submitted 2022-03-03; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Myocarditis and Cardiomyopathy
Keywords: SARS CoV-19; Vaccination
MeSH Terms: conditions — Myocarditis; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background The novel coronavirus disease 2019 (COVID-19) caused by an infection with the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has rapidly become a global pandemic with more than 190.000.000 infections and 4.250.000 reported deaths worldwide.

SARS-CoV-2 vaccination plays an important role in containing the pandemic and the possible adverse complications of COVID-19. Large clinical trials have proven the safety and efficacy of the vaccines currently in use. Systemic reactions usually were mild, self-limiting and could be observed more often in younger vaccine recipients. Cases of myocarditis after vaccination have been reported for various vaccines. The new vaccines for SARS-CoV-2 also seem to be affected by this adverse reactions. The pathophysiology is uncertain so far.

Aim Aim of this study is a systematic registration of myocarditis cases associated with SARS-CoV-2 vaccination which were diagnosed and/or treated in participating centers. The main goal of this study is the characterization of clinical manifestations and prognosis of the disease.

Study Design Patient history, laboratory tests and cardiovascular imaging data of patients with suspected SARS-CoV-2 - vaccine associated myocarditis are documented. Patients with clinical suspicion of troponin-positive myocarditis within 30 days after receiving SARS-CoV-2 vaccine without evidence for apparent other causes e.g. infectious or autoimmune etiology were included. Clinical follow-up data is acquired.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 Vaccine-associated Myocarditis (< 30 days after vaccination) confirmed by cardiac MRI without evidence of alternative etiology (infectious, auto-immune myocarditis).

Exclusion Criteria:

* missing individual consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with SARS-CoV-2 Vaccine-associated Myocarditis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Combined Primary Endpoint | 6 months
  Death, Hospitalization, symptomatic Heart Failure

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ochs, MD, Principal Investigator — Theresien Hospital Mannheim
Locations (1):
- Theresienkrankenhaus, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schroth D, Garg R, Bocova X, Hansmann J, Haass M, Yan A, Fernando C, Chacko B, Oikonomou A, White J, Alhussein MM, Giusca S, Ochs A, Korosoglou G, Andre F, Friedrich MG, Ochs M. Predictors of persistent symptoms after mRNA SARS-CoV-2 vaccine-related myocarditis (myovacc registry). Front Cardiovasc Med. 2023 Jun 21;10:1204232. doi: 10.3389/fcvm.2023.1204232. eCollection 2023. PMID 37416926